CLINICAL TRIAL: NCT01353794
Title: Prospective, Multicentric, Large Scale Observational Study to Evaluate Effectiveness and Safety of Nexavar® in Advanced Renal Cell Carcinoma
Brief Title: Study to Observe Safety and Efficacy of Nexavar in Treatment of Kidney Cancer
Acronym: POWER-NEXT
Status: Withdrawn | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 15246; NX0913IN (Other: Company Internal)
Record Dates: First submitted 2011-05-13; First posted 2011-05-16 (Estimated); Last update posted 2015-01-30 (Estimated); Status verified 2015-01

CONDITIONS: Carcinoma, Renal Cell
Keywords: SORAFENIB; RENAL CELL CARCINOMA; TYROSINE KINASE INHIBITOR; OBSERVATIONAL STUDY
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — The treatment with Sorafenib 200mg tablets should comply with the recommendations written in the local product information. The decision about the duration of treatment is solely at the discretion of the attending physician

SUMMARY:
The objective of this Non-Interventional study is to evaluate the effectiveness & safety of Nexavar in advanced Renal Cell Carcinoma (RCC) patients under daily-life treatment conditions based on age of the patient (older (age >70 years) and younger patients (age <70 years). Specifically investigated are the tumor status, duration of Nexavar ® treatment (number of cycles) and incidence of Hand foot Skin Reaction.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of advanced Renal Cell Carcinoma (RCC) and decision taken by the investigator to prescribe Sorafenib

Exclusion Criteria:

* Exclusion criteria must be read in conjunction with the local product information.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients of advanced RCC
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-12; Primary Completion 2017-09 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Efficacy related variables are status of tumor / metastases. | After 12 months, or at discontinuation of therapy or at end of study (whatever is earlier)
Efficacy related variables are patient's performance status. | After 12 months, or at discontinuation of therapy or at end of study (whatever is earlier)
Efficacy related variables are efficacy assessment by the physician. | After 12 months, or at discontinuation of therapy or at end of study (whatever is earlier)
Efficacy related variable - Quality of Life (QOL) assessment by the patient | After 12 months, or at discontinuation of therapy or at end of study (whatever is earlier)

SECONDARY OUTCOMES:
General tolerability assessment by physician and reports of adverse events. | After 12 months, or at discontinuation of therapy or at end of study (whatever is earlier)

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer